CLINICAL TRIAL: NCT02488369
Title: Study on the Diagnostic Qualities of the Positron Emission Tomography Coupled to the Scanner (PET / CT) in the Assessment of Response to Non-Hodgkin's Lymphoma Therapy in Children and Adolescents
Brief Title: Diagnostic Qualities of the Positron Emission Tomography Coupled to the Scanner (PET / CT) in the Assessment of Response to Non-Hodgkin's Lymphoma Therapy in Children and Adolescents
Acronym: TEP-LYMPHOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Société Française des Cancers et Leucémies de l'Enfant et de l'Adolescent (SFCE) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010-A01154-35; 2010/1651 (Other: CSET number)
Record Dates: First submitted 2015-06-29; First posted 2015-07-02 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: Children and adolescents
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with non-Hodgkin's lymphoma (Experimental)
  Interventions: Device: PET / CT

INTERVENTIONS:
Device: PET / CT

SUMMARY:
This is a diagnostic prospective multicenter study. This study will be conducted in 32 centers of the Société Française des Cancers et Leucémies de l'Enfants et de l'Adolescent (SCFE) in patients with non-Hodgkin lymphoma and treated according to recommendations of the SFCE for each type of non-Hodgkin lymphoma. All patients will have a PET / CT associated with conventional imaging time of remission assessment. Histological examination of residual tumor will be conducted whenever practicable in patients with pathologic residual image on conventional imaging and / or PET / CT. A central review of conventional imaging examinations and PET / CT will be performed independently from each other.

Moreover, whenever possible, patients will have a PET / CT at diagnosis and an early PET / CT (between J8 and J28 according to the type of lymphoma and toxicities due to treatment). The results of the early PET / CT should not lead to treatment modifications.

In case of residual tumor at remission assessment, therapeutics changes as recommended therapeutic protocols will be based on histologic findings and not on the results of PET / CT alone.

ELIGIBILITY:
Inclusion Criteria:

1. All cases of NHL corresponding to one of the following histologies:

   * Burkitt and Burkitt-like (LB)
   * Large cell B-cell lymphoma (LBGC)
   * Primary mediastinal B cell lymphoma (LBPM)
   * Lymphoblastic lymphoma (LL)
   * Anaplastic large cell lymphoma (ALCL)
2. Age > 2 years and < 21 years
3. Treated in a SFCE protocol
4. Treated in a center with the possibility of organizing a PET / CT at the time of remission assessment
5. Affiliation to a social security system
6. Possible follow-up for at least 2 years
7. written informed consent signed by the parents or parental authority or the patient himself if he is over 18 years

Exclusion Criteria:

1. relapsing patients
2. Patients with absolute cons-indications to the achievement of a PET scan: pregnancy, incontinence, poorly controlled diabetes or blood glucose> 10 mmol/l, alterations of superior functions or claustrophobia, making the test impossible.
3. pre-existing or evolving infectious inflammatory disease making PET / CT difficult to interpret

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 230 (Actual)
Dates: Start 2011-03-31 (Actual); Primary Completion 2015-08-03 (Actual); Study Completion 2018-01-25 (Actual)

PRIMARY OUTCOMES:
PET sensitivity according to Juweid et Cheson criterias | 28 days after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy Cancer Campus Grand Paris, Villejuif, Val De Marne, France